CLINICAL TRIAL: NCT06123260
Title: Short Term Renal Outcomes Among Post Liver Transplantation Patients at Assiut University
Brief Title: Renal Outcomes Among Post Liver Transplantation Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ebram Magdy Eskander Nashed, doctor, Assiut University
Other Study IDs: renal outcomes post OLT
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Liver Transplant; Complications; Renal Complication of Procedure
MeSH Terms: interventions — Kidney Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: renal function tests — BUN, eGFR , CBC , Electrolytes , Liver function tests

SUMMARY:
To evaluate Renal outcomes among patients, post liver transplantation at Assiut university.

DETAILED DESCRIPTION:
It is estimated that 1 in 4 liver transplantation (LT) recipients has an estimated glomerular filtration rate (eGFR) of <60mL/minute/1.73 m2 at the time of LT Renal dysfunction, both before or after LT, is an important comorbidity associated with an increased risk of death, morbidity, and cost. Serum creatinine, a major component of the Model for End-Stage Liver Disease (MELD) score, has driven the increased incidence of renal dysfunction among patients undergoing LT End-stage liver disease (ESLD) is commonly complicated by kidney dysfunction, which in turn leads to a worse prognosis. The kidney dysfunction can be functional or structural, ranging from prerenal azotemia and hepatorenal syndrome causing acute kidney injury to immunoglobulin A (IgA) nephropathy (IgAN) and membranoproliferative glomerulonephritis causing chronic kidney disease Each condition carries a different presentation, treatment, prognosis, and risk of recurrence. Therefore, when ESLD patients undergo evaluation for liver transplant, it is critical to assess their kidney function and understand the cause of any underlying kidney dysfunction LT recipients will continue to worsen due to calcineurin inhibitor toxicity and lack of recovery from hepatorenal syndrome (HRS), necessitating renal replacement therapy Patients who are not expected to recover their kidney function after liver transplant usually benefit from combined liver and kidney transplant (CLKT). Others may need modified immunosuppressive regimens that minimize or avoid use of calcineurin inhibitors to preserve the remaining kidney function.

For assessment of kidney function, Equations that estimate GFR are most commonly used in daily practice. They have the advantage of being inexpensive and results are immediately available. Their disadvantage is that they rely on endogenous biomarkers, which are confounded by non-GFR determinants such as age, sex, muscle mass, drugs, certain chronic conditions, diet and presumably many more Creatinine, the most commonly used biomarker, depends heavily on muscle mass. Pre and intraoperative factors and postoperative complications were evaluated for their impact on development of AKI The preoperative factors MELD, SCr, Bilirubin and INR were highly associated with an increased risk for developing AKI requiring RRT for the post OLT complications, length of ICU stay was associated with the development of AKI Patients with a longer ventilation time and a higher amount of RPC transfusion were more likely to have AKI requiring RRT, whereas these parameters were not associated with milder forms of AKI.

ELIGIBILITY:
Inclusion Criteria:

* Data of all Patients underwent liver transplants with their reports available at El Raghy university hospital

Exclusion Criteria:

* Inadequate data
* Patients on dialysis more than 8 weeks pre liver transplant.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: retrospective cohort study will be done to patients post liver transplantation at El Raghy university hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
calculation the incidence of AKI in Liver transplantation patients | Baseline
  Determination of the most common risk factor for AKI in liver transplantation patients.

SECONDARY OUTCOMES:
mortality rate | Baseline
  patient survival in post LT AKI group.

CONTACTS AND LOCATIONS:
Overall Officials: Bahaa Osman Taha, Master, Study Director — Bahaa_osman99@aun.edu.eg

REFERENCES:
- [Background] Feffer SE, Parray HR, Westring DW. Seizure after infusion of aminocaproic acid. JAMA. 1978 Nov 24;240(22):2468. No abstract available. PMID 101682
- [Background] Rautela GS, Snee RD, Miller WK. Response-surface co-optimization of reaction conditions in clinical chemical methods. Clin Chem. 1979 Nov;25(11):1954-64. PMID 498506
- [Background] Ramakrishnan R, Mittal S, Ambatkar S, Kader MA. Retinal nerve fibre layer thickness measurements in normal Indian population by optical coherence tomography. Indian J Ophthalmol. 2006 Mar;54(1):11-5. doi: 10.4103/0301-4738.21608. PMID 16531664
- [Background] Braun OH, Kreipe U. [Rare forms of chronic osteomyelitis in children (author's transl)]. Klin Padiatr. 1979 Sep;191(5):511-21. German. PMID 574584
- [Background] Pannuti F. Surgical adjuvant hormone therapy in breast cancer. Arch Geschwulstforsch. 1978;48(7):680-2. No abstract available. PMID 736749
- [Background] Pozenel H. [The influence of mexiletin on ventricular arrhythmias during ergometric exercise (author's transl)]. Wien Klin Wochenschr. 1977 Dec 9;89(23):783-8. German. PMID 595602
- [Background] Blom E. A decapitated sperm defect in two sterile Hereford bulls. Nord Vet Med. 1977 Mar;29(3):119-23. PMID 870880